CLINICAL TRIAL: NCT04326907
Title: Efficacy and Safety of Treatment of Complex Anal Fistulas Not Associated With Crohn's Disease Using Centrifuged Adipose Tissue Containing Progenitor Cells: a Randomized Controlled Clinical Trial
Brief Title: Treatment of Complex Anal Fistulas Using Centrifuged Adipose Tissue Containing Progenitor Cells
Acronym: CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Simona Ascanelli, Principal Investigator, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHFerrara160597
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Anal Fistula
Keywords: complex fistula-in ano; adipose tissue; stem cell therapy
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: This monocentric randomized controlled study was designed to test the efficacy and safety of injection of CAT for treatment of complex fistula-in ano, not associated with CD . Eligible patients were randomly assigned, according to a 1:1 scheme, to receive treatment with or without CAT. In the experimental arm, anal fistulas were treated by conventional surgery, and CAT injection. No experimental treatment (CAT) was administered to the control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- CAT injection group (Experimental): After fistulectomy for complex anal fistula, CAT (harvested from abdominal subcutaneous adipose tissue by Coleman's procedure) was injected into the tissue surrounding the internal opening, and inside the perianal wound obtained after fistulectomy.
  Interventions: Procedure: Autologous centrifuged adipose tissue (CAT) injection after anal fistulectomy
- No CAT injection group (No Intervention): Patients of this group were treated with anal fistulectomy without CAT injection.

INTERVENTIONS:
Procedure: Autologous centrifuged adipose tissue (CAT) injection after anal fistulectomy — Collection and injection of autologous adipose tissue in complex anal fistulas in one surgical step under locoregional or general anesthesia.
  Arms: CAT injection group

SUMMARY:
In the treatment of complex anal fistulas transplant of freshly collected autologous adipose tissue mechanically fragmented or centrifuged adipose tissue (CAT) might be an alternative to in vitro expanded autologous or allogeneic adipose-derived stem cells, showing remarkable efficacy in diverse therapeutic indications.

The aim of our study is to evaluate randomly the efficacy and safety of the use of CAT in the healing process of complex anal fistulas, except for Crohn's disease (CD) related fistulas.

DETAILED DESCRIPTION:
This monocentric randomized controlled study was designed to test the efficacy and safety of injection of CAT for treatment of complex fistula-in ano, not associated with CD . The study was conducted at the Second Surgical Unit of the University Hospital of Ferrara, located in the North East of Italy. All consecutive patients referred to our clinic with complex anal fistula were screened. Patients were enrolled from May 2016 through May 2019.

Eligible patients were randomly assigned, according to a 1:1 scheme, to receive treatment with or without CAT (120 patients totally). The primary endpoint was defined as the proportion of patients whose fistula was completely healed within 4 weeks after surgery. Fistula healing was defined as the absence of any anal symptom, with no discharge from the fistula and a closed external opening confirmed on clinical evaluation. Fistula healing was eventually confirmed by a pelvic MRI at 3 months after surgery.Moreover, we analyzed postoperative pain measured by Visual Analogue Scale for 2 weeks after surgery to evaluate whether CAT injection could modulate pain, and recurrence at 6 months to evaluate the long-term efficacy of CAT injection.

Faecal continence was assessed before surgery and at 6-months follow-up visit using the Cleveland Clinical Florida Fecal Incontinence (CCF-FI) questionnaire. Adipose tissue from periombelical or lateral abdomen was harvested from these patients by liposuction to prepare CAT using Coleman's technique.Complex anal fistulas were treated by conventional surgery. Once the seton (present in the most of patients) was removed, after identification of internal opening, necrotic and inflamed tissues were excised using a "cone-like" fistulectomy or debrided with a wire brush to remove granulation tissue by the help of fistuloscope (VAAFT modified, without destroying the fistulous track with monopolar electrode). Before CAT injection, the internal opening was treated in two ways: by simply closing it using 2-0 Vicryl stitches on the muscular and mucosal layers or by performing a mucosal advancement rectal flap.

CAT was injected into the submucosal layer surrounding the internal opening, and around the fistula tract wall (in case of VAAFT modified) or inside the perianal wound after fistulectomy, using a 1-mL syringe equipped with a 22-gauge and 30-mm length needle, dividing injections at all quadrants of fistula wall, or distributing the CAT inside the perianal wound, at different levels by using multiple passes from the internal to the external openings until there was firm swelling surrounded the fistula tract. The external opening was approximated loosely with a suture to allow drainage of the fistula, but not extrusion of the centrifuged adipose tissue. The amount of product injected may vary depending on the total amount harvested but it should be not less than 10 ml. Patients were assessed for fistula healing, pain (VAS) and AEs at 1 week, 2 weeks, 4 weeks, 8 weeks, three months, and 6 months after treatment. Assessment consisted of clinical examination and AEs and VAS registration. Pelvic MRI was performed at 3 months after surgery. The Cleveland Clinical Florida Fecal Incontinence (CCF-FI) questionnaire was administered before surgery and at 6-months follow-up visit. At the final visit patients were also asked about their overall satisfaction with the procedure, with ratings from very satisfied to very dissatisfied.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or older with complex perianal fistulas

Exclusion Criteria:

Inflammatory bowel diseases, Crohn's Disease (CD) or Ulcerative Colitis (UC) Hepatitis B or C virus Infection with Human immunodeficiency virus Surgery for a malignant tumor during the previous 5 years (excluding in situ carcinoma) Previous pelvic radiotherapy Autoimmune disease Active tuberculosis Symptoms of septicemia Breastfeeding or pregnant women Women unwilling to use contraception during the study Psychiatric disorders Alcoholism Drug dependency Allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Fistula healing rate within 6 months after surgery | up to 6 months
  Fistula healing was defined as the absence of any anal symptom, with no discharge from the fistula and a closed external opening confirmed on clinical evaluation. Fistula healing was eventually confirmed by a pelvic MRI at 3 months after surgery

SECONDARY OUTCOMES:
Safety of autologous adipose tissue injection | 4 weeks
  Safety was evaluated by the overall incidence and severity of Adverse Events (AEs) up to 4 weeks following surgery.

OTHER OUTCOMES:
postoperative pain | 2 weeks
  postoperative pain measured by Visual Analogue Scale (0-10) for 2 weeks after surgery to evaluate whether CAT injection could modulate pain
recurrence at 6 months | 6 months
  to evaluate the long-term efficacy of CAT injection

CONTACTS AND LOCATIONS:
Overall Officials: Simona Ascanelli, MD, Principal Investigator — University Hospital Ferrara
Locations (1):
- Simona Ascanelli, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data access requests will be reviewed by an external indipendent review Panel. Requestores will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Limura E, Giordano P. Modern management of anal fistula. World J Gastroenterol. 2015 Jan 7;21(1):12-20. doi: 10.3748/wjg.v21.i1.12. PMID 25574077
- [Result] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Result] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960
- [Result] Aust L, Devlin B, Foster SJ, Halvorsen YD, Hicok K, du Laney T, Sen A, Willingmyre GD, Gimble JM. Yield of human adipose-derived adult stem cells from liposuction aspirates. Cytotherapy. 2004;6(1):7-14. doi: 10.1080/14653240310004539. PMID 14985162
- [Result] Zuk PA, Zhu M, Ashjian P, De Ugarte DA, Huang JI, Mizuno H, Alfonso ZC, Fraser JK, Benhaim P, Hedrick MH. Human adipose tissue is a source of multipotent stem cells. Mol Biol Cell. 2002 Dec;13(12):4279-95. doi: 10.1091/mbc.e02-02-0105. PMID 12475952
- [Result] Naldini G, Sturiale A, Fabiani B, Giani I, Menconi C. Micro-fragmented adipose tissue injection for the treatment of complex anal fistula: a pilot study accessing safety and feasibility. Tech Coloproctol. 2018 Feb;22(2):107-113. doi: 10.1007/s10151-018-1755-8. Epub 2018 Feb 16. PMID 29453515
- [Result] Dige A, Hougaard HT, Agnholt J, Pedersen BG, Tencerova M, Kassem M, Krogh K, Lundby L. Efficacy of Injection of Freshly Collected Autologous Adipose Tissue Into Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2019 Jun;156(8):2208-2216.e1. doi: 10.1053/j.gastro.2019.02.005. Epub 2019 Feb 14. PMID 30772343
- [Result] Laureti S, Gionchetti P, Cappelli A, Vittori L, Contedini F, Rizzello F, Golfieri R, Campieri M, Poggioli G. Refractory Complex Crohn's Perianal Fistulas: A Role for Autologous Microfragmented Adipose Tissue Injection. Inflamm Bowel Dis. 2020 Jan 6;26(2):321-330. doi: 10.1093/ibd/izz051. PMID 31220252
- [Result] Pu LLQ, Coleman SR, Cui X, Ferguson REH Jr, Vasconez HC. Autologous fat grafts harvested and refined by the Coleman technique: a comparative study. Plast Reconstr Surg. 2008 Sep;122(3):932-937. doi: 10.1097/PRS.0b013e3181811ff0. PMID 18766062
- [Result] Ibatici A, Caviggioli F, Valeriano V, Quirici N, Sessarego N, Lisa A, Klinger F, Forcellini D, Maione L, Klinger M. Comparison of cell number, viability, phenotypic profile, clonogenic, and proliferative potential of adipose-derived stem cell populations between centrifuged and noncentrifuged fat. Aesthetic Plast Surg. 2014 Oct;38(5):985-93. doi: 10.1007/s00266-014-0372-9. Epub 2014 Jul 23. PMID 25053112
- [Result] Zollino I, Campioni D, Sibilla MG, Tessari M, Malagoni AM, Zamboni P. A phase II randomized clinical trial for the treatment of recalcitrant chronic leg ulcers using centrifuged adipose tissue containing progenitor cells. Cytotherapy. 2019 Feb;21(2):200-211. doi: 10.1016/j.jcyt.2018.10.012. Epub 2018 Dec 22. PMID 30583949
- [Result] Park SR, Kim JW, Jun HS, Roh JY, Lee HY, Hong IS. Stem Cell Secretome and Its Effect on Cellular Mechanisms Relevant to Wound Healing. Mol Ther. 2018 Feb 7;26(2):606-617. doi: 10.1016/j.ymthe.2017.09.023. Epub 2017 Oct 5. PMID 29066165
- [Result] Vezzani B, Shaw I, Lesme H, Yong L, Khan N, Tremolada C, Peault B. Higher Pericyte Content and Secretory Activity of Microfragmented Human Adipose Tissue Compared to Enzymatically Derived Stromal Vascular Fraction. Stem Cells Transl Med. 2018 Dec;7(12):876-886. doi: 10.1002/sctm.18-0051. Epub 2018 Sep 26. PMID 30255987
- [Derived] Ascanelli S, Zamboni P, Campioni D, Grazia Sibilla M, Chimisso L, Zollino I, Valpiani G, Carcoforo P. Efficacy and Safety of Treatment of Complex Idiopathic Fistula-in-Ano Using Autologous Centrifuged Adipose Tissue Containing Progenitor Cells: A Randomized Controlled Trial. Dis Colon Rectum. 2021 Oct 1;64(10):1276-1285. doi: 10.1097/DCR.0000000000001924. PMID 34016825